CLINICAL TRIAL: NCT02015182
Title: Bupivacaine Pharmacokinetics in Children Following Transversus Abdominis Plane Block
Brief Title: Bupivacaine Pharmacokinetics Following TAP Block
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Jason Hayes, Staff Anesthesiologist, The Hospital for Sick Children
Other Study IDs: 1000023222
Record Dates: First submitted 2013-08-21; First posted 2013-12-19 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Transversus Abdominis Plane Block
Keywords: Bupivacaine; Sensorcaine; Population pharmacokinetics; Children; Pediatrics; Transversus abdominis plane (TAP) block; Regional Anesthesia
MeSH Terms: conditions — Bites and Stings | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood (serum)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Blood sample for bupivicaine pharmacokinetics: Children undergoing TAP block will have blood sampled for bupivacaine pharmacokinetics
  Interventions: Other: Blood sample for bupivicaine pharmacokinetics

INTERVENTIONS:
Other: Blood sample for bupivicaine pharmacokinetics — Bupivacaine levels will be measured with an assay developed on the 4000 QTrap Tandem Mass Spectrometer (Applied Biosystems/ MDS Sciex).
  Data will be collected and analyzed using the Agilent ChemStation software (Rev A.10.02). The analytical column is an Agilent Zorbax Eclipse XDB-C8 (4.6 x 150mm, 5µm).Quantification of bupivacaine is based on analyzing a six point calibration curve (0 to 4.0 mg/L). An internal standard (Prilocaine 221.2/86.1) is included with each calibrator, quality control or patient sample. Instrumentation and Chromatographic conditions: The HPLC system consists of a Specta-System P1000 Isocratic Pump and an AS3000 Autosampler (Thermo Electron Corporation, Waltham MA).

SUMMARY:
The aims of this study are to determine population PK parameters of bupivacaine in children following TAP block using a population-based PK approach, and to evaluate the influence of patient covariates on drug disposition.

DETAILED DESCRIPTION:
The number of published pediatric studies on the use of transversus abdominis plane (TAP) block has increased in recent years. The transversus abdominis plane (TAP) block has been used for postoperative analgesia for surgery to the abdominal wall and involves the injection of local anesthetic solution into a plane between internal oblique (IO) and transversus abdominis (TA) muscles. The TAP block has the advantage of providing unilateral analgesia in instances of non-midline abdominal incision and is particularly useful in cases where epidural blockade is either contraindicated or technically or logistically not feasible. Bupivacaine and ropivacaine have been used as local anesthetics for TAP blocks in published studies to date. However, no data exist regarding the pharmacokinetics of bupivacaine after TAP block in children. The aims of this study are to determine population pharmacokinetic (PK) parameters of bupivacaine in children following a TAP block, using a population-based PK approach.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving a TAP block as part of routine anesthetic management
* Patients older than 3 months and less than 18 years of age
* Patients weighing ≥ 6 kg
* Patients with American Society of Anesthesiologists (ASA) score 1-3

Exclusion Criteria:

* Patients with known severe preexisting liver disease
* Patients with known severe (i.e. requiring dialysis) preexisting renal disease
* Patients who will be discharged the day of surgery
* Refusal to consent

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children undergoing TAP block for postoperative pain control
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Population pharmacokinetics of bupivacaine and the influence of patient covariates on drug disposition | 0 - 360 minutes after the TAP block is performed
  Blood will be drawn from an indwelling intravenous catheter. Each patient will have a total of 6 samples collected during each of the following time blocks: 0 - 10 minutes, 11 - 20 minutes, 21 - 30 minutes, 31 - 60 minutes, 61 - 180 minutes and 181 - 360 minutes after the TAP block is performed. Age, weight, sex, concomitant drugs (intravenous and inhalation anesthetics, muscle relaxants, and opioids), and kidney function data will be investigated as co-variables for each of the primary parameters. We will obtain estimates of total clearance (CL), volume of distribution, elimination half life (t1/2), estimates of clearance, and absorption rate constant.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Hayes, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada